CLINICAL TRIAL: NCT06788327
Title: Comparing the Effectiveness of Blood Flow Restriction Therapy Versus Standard Exercise After Arthroscopic Rotator Cuff Repair: Protocol for the Multicenter S-TRONGER Randomized Controlled Trial
Brief Title: Blood Flow Restriction Versus Standard Exercise After Rotator Cuff Repair
Acronym: S-TRONGER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, José Casaña Granell, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BFRT in RCR rehabilitation
Record Dates: First submitted 2025-01-15; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Rotator Cuff Injury; Rotator Cuff Tears; Rotator Cuff Repair
Keywords: blood flow restriction therapy; blood flow restriction training
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Opaque sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard exercises with BFRT (Experimental): Participants with arthroscopic rotator cuff repair will undergo rehabilitation using progressive exercises with BFRT during the three phases of standard rehabilitation.
  Interventions: Other: Standard rehabilitation; Device: Blood Flow Restriction Therapy
- Standard exercises alone (Active Comparator): Participants with arthroscopic rotator cuff repair will undergo rehabilitation using progressive exercises without BFRT during the three phases of standard rehabilitation.
  Interventions: Other: Standard rehabilitation

INTERVENTIONS:
Other: Standard rehabilitation — Protocol based on the best available evidence and to be used in all participants in both groups. The standard exercises protocol will consist of three postoperative rehabilitation phases: phase I (weeks 1 to 4), phase II (weeks 5 to 8) and phase III (weeks 9 to 12). Sessions will be held 2 times a week for 12 weeks. Each session will last 45 minutes and will consist of six exercises in the phase I, eight exercises in phase II, and eight exercises in phase III.
Device: Blood Flow Restriction Therapy — Participants will perform three exercises of the standard exercises protocol with BFRT. An auto-regulated portable BFRT SmartCuffs® 3.0 Pro system with a 17-inch long and 5-inch-wide cuff (Smart Tools Plus, United States), placed on the most proximal part of the arm, will be used. Each BFRT session will begin with a maximal occlusion test to personalize the occlusion pressure to the participant. The limb occlusion pressure (LOP) will be set at 50% of the maximum occlusion pressure in the first stage and 60% in stages II and III. The participant will perform 75 repetitions per BFRT exercise divided into 4 sets (30, 15, 15, and 15 repetitions). The load intensity during the BFRT exercises will be set near to 3 out of 10 on the Borg's CR10 scale ("weak"), which corresponds to 30% of a 1RM effort. After each exercise, the cuff will be deflated, and the patient will rest for two minutes.
  Arms: Standard exercises with BFRT

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of postoperative standard exercises with blood flow restriction therapy (BFRT) versus standard exercises alone on shoulder muscle strength and mass in participants with surgically treated rotator cuff tear. It is presumed that the addition of BFRT will significantly improve the shoulder strength and muscle mass at the end of the intervention period compared to the group receiving only standard exercises.

Patients who agree to participate in this research will be randomly assigned to a control group (standard exercises alone) or an experimental group (standard rehabilitation with BFRT). The duration of the postoperative intervention will be 12 weeks. The primary variables will be the shoulder muscle strength and muscle mass. Secondary variables will be the active shoulder mobility, pain intensity, upper limb disability, and health-related quality of life. Results will be measured at 0, 4 and 12 weeks postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-65 years
* Symptomatic degenerative rotator cuff tear diagnosed by magnetic resonance imaging
* Undergoing arthroscopic rotator cuff repair
* Be able to read and understand Spanish

Exclusion Criteria:

* Massive irreparable rotator cuff tear
* Concomitant fracture
* Labral or nerve injury
* Suspicious of developing a frozen shoulder
* Revision surgery after rotator cuff repair
* Previous corticosteroid injection (< 6 months)
* Recent surgery (< 1 year) in the contralateral shoulder
* History of deep venous thrombosis/pulmonary embolism, peripheral vascular disease, thrombophilia or clotting disorders
* Severe or uncontrolled hypertension, or any comorbid condition that impedes participants to complete the intervention

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder muscle strength | 0, 4 and 12 weeks
  Shoulder abduction and external rotation maximum voluntary isometric strength will be measured using dynamometry (kilograms)
Shoulder muscle mass | 0, 4 and 12 weeks
  Supraspinatus and long head biceps brachii tendon thickness will be measured using ultrasound imaging (milimeters)

SECONDARY OUTCOMES:
Active Range of Motion | 0, 4 and 12 weeks
  Shoulder flexion, abduction, and external rotation will be measured with a goniometer (degrees)
Pain intensity | 0, 4 and 12 weeks
  Visual Analogue Scale (0 to 10 centimeters)
Self-reported upper limb disability | 0, 4 and 12 weeks
  Shoulder Pain Disability Index (0 to 100%)
Self-reported quality of life | 0, 4 and 12 weeks
  Western Ontario Rotator Cuff Index (0 to 100%)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Ponce-Fuentes, MSc, Principal Investigator — Universidad Mayor
Locations (1):
- Clínica RedSalud Mayor, Temuco, Cautín, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Background] Lambert BS, Hedt C, Ankersen JP, Goble H, Taft C, Daum J, Karasch R, Moreno MR, McCulloch PC. Rotator cuff training with upper extremity blood flow restriction produces favorable adaptations in division IA collegiate pitchers: a randomized trial. J Shoulder Elbow Surg. 2023 Jun;32(6):e279-e292. doi: 10.1016/j.jse.2023.02.116. Epub 2023 Mar 17. PMID 36933646
- [Background] Lambert B, Hedt C, Daum J, Taft C, Chaliki K, Epner E, McCulloch P. Blood Flow Restriction Training for the Shoulder: A Case for Proximal Benefit. Am J Sports Med. 2021 Aug;49(10):2716-2728. doi: 10.1177/03635465211017524. Epub 2021 Jun 10. PMID 34110960
- [Background] Kjaer BH, Magnusson SP, Henriksen M, Warming S, Boyle E, Krogsgaard MR, Al-Hamdani A, Juul-Kristensen B. Effects of 12 Weeks of Progressive Early Active Exercise Therapy After Surgical Rotator Cuff Repair: 12 Weeks and 1-Year Results From the CUT-N-MOVE Randomized Controlled Trial. Am J Sports Med. 2021 Feb;49(2):321-331. doi: 10.1177/0363546520983823. Epub 2021 Jan 20. PMID 33471547
- [Background] Kara D, Ozcakar L, Demirci S, Huri G, Duzgun I. Blood Flow Restriction Training in Patients With Rotator Cuff Tendinopathy: A Randomized, Assessor-Blinded, Controlled Trial. Clin J Sport Med. 2024 Jan 1;34(1):10-16. doi: 10.1097/JSM.0000000000001191. Epub 2023 Sep 14. PMID 37706671
- [Background] Hughes L, Patterson SD. The effect of blood flow restriction exercise on exercise-induced hypoalgesia and endogenous opioid and endocannabinoid mechanisms of pain modulation. J Appl Physiol (1985). 2020 Apr 1;128(4):914-924. doi: 10.1152/japplphysiol.00768.2019. Epub 2020 Feb 27. PMID 32105522
- [Background] Bowman EN, Elshaar R, Milligan H, Jue G, Mohr K, Brown P, Watanabe DM, Limpisvasti O. Upper-extremity blood flow restriction: the proximal, distal, and contralateral effects-a randomized controlled trial. J Shoulder Elbow Surg. 2020 Jun;29(6):1267-1274. doi: 10.1016/j.jse.2020.02.003. PMID 32423577
- See also: Ponce-Fuentes, F., Cuyul-Vásquez, I., Carranza, J., Lluch, E., Calatayud, J., Casaña, J., ... & Struyf, F. (2024). Early Rehabilitation With Blood Flow Restriction Therapy Following Arthroscopic Rotator Cuff Repair: A Case Report. JOSPT Cases, 4(3) — https://www.jospt.org/doi/abs/10.2519/josptcases.2024.0052